CLINICAL TRIAL: NCT02199405
Title: Study on the Early Warning and Treatment of Cervical Spondylosis of Cervical Type on Young People Based on the " Move Generate Yang " Theory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wang Yucheng (Other)
Responsible Party: Sponsor-Investigator, Wang Yucheng, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Organization: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13066
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Cervical Spondylosis of Cervical Type
Keywords: Spondylosis, Massage Therapy, Exercise Therapy ,Treatment Efficacy
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- massage and Sishi Daoyin (Experimental): Massage of chiropractic and adjusting cervical curvature, 10 minutes, three times one week for 4 weeks Sishi Daoyin, practicing during 9-11am, once a day for 4 weeks
  Interventions: Other: Massage of chiropractic and adjusting cervical curvature; Other: Sishi Daoyin
- conventional massage and cervical traction (Active Comparator): Conventional massage , 15 minutes, three times one week for 4 weeks Cervical traction , 15 minutes, three times one week for 4 weeks
  Interventions: Other: conventional massage; Other: Cervical traction

INTERVENTIONS:
Other: Massage of chiropractic and adjusting cervical curvature — Massage of chiropractic and adjusting cervical curvature, 10 minutes, three times one week for 4 weeks
  Arms: massage and Sishi Daoyin
Other: Sishi Daoyin — Sishi Daoyin, practicing during 9-11am, once a day for 4 weeks
  Arms: massage and Sishi Daoyin
Other: conventional massage — Conventional massage , 15 minutes, three times one week for 4 weeks
  Arms: conventional massage and cervical traction
Other: Cervical traction
  Other Names: Cervical traction , 15 minutes, three times one week for 4 weeks
  Arms: conventional massage and cervical traction

SUMMARY:
The incidence of cervical spondylosis on young people is increasing every year. Suffering from this disease will affect the normal life and learning of young people. Episode younger and incidence higher of this disease could increase health care spending of the government in the economy. Cervical spondylosis of cervical type is the main type of cervical spondylosis of young people. Patients of cervical spondylosis of cervical type always manifest the head, neck and shoulder pain accompanied by corresponding pressure point, the X-ray display of Upper cervical curvature change and instability of intervertebral joint performance ,and the dynamic lateral X-ray shows vertebral instability or trapezoidal change. The conservative treatment is the primary and preferred treatment of the disease.

This study is designed as a random, control, single blind study. It will recruit 140 cases of cervical spondylosis of cervical type. Both the treatment group and the control group will be randomly assigned 70 cases. Patients in the treatment group will be treated by Massage of chiropractic and adjusting cervical curvature and practice Sishi Daoyin for 4 weeks，and the control group by conventional massage and cervical traction. The total study includes 2 views that are baseline and post-4week intervention. At all of the 2 views, all participants will be examined range of motion of cervical vertebra, cervical curvature, and Surface Electromyography of neck muscles, and will be estimated scores of The Neck Disability Index(NDI), the Northwick Park Neck Pain Questionnaire (NPQ),Short-form McGill Pain Questionnaire(SF-MPQ) and Evaluation of the therapeutic effect. This study aims to investigate the efficacy of Massage of chiropractic and adjusting cervical curvature and Sishi Daoyin practice, and discover the correlation between these scales and these objective indicators to discover the indicators of early warning signs of cervical spondylosis of cervical type of young people.

DETAILED DESCRIPTION:
Quality control: The study site and all researchers must comply with the required qualifications. All researchers must be trained before the study. The study will take a number of measures to ensure the recruitment of the required sample size, and compliance of intervention providers and participants.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria of cervical spondylosis of cervical type
* first invasion and not receive any treatment
* X-ray shows cervical curvature go straight
* volunteered to join the test, and sign " informed consent " persons

Exclusion Criteria:

* suspected or confirmed bone and joint and soft tissue tumors, and so on
* suffer from cardiovascular, lung, liver, kidney and hematopoietic system serious illness or impairment
* lesions of skin ( such as damage, burns, and so on ) where massage will be applied
* severe congenital malformation of cervical vertebra
* incapacitated or unable to independently read and write
* other conditions which researchers consider appropriate to participate in this study

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
value of cervical curvature | baseline and post- 4week intervention
  We will examine the value of cervical curvature of participants at baseline and post- 4week intervention.

SECONDARY OUTCOMES:
range of motion of cervical vertebra | baseline and post- 4week intervention
  We will examine the range of motion of cervical vertebra, including cervical flexion, extension, flexion to the left, flexion to the right, rotation to the left and rotation to the right.
value of Surface Electromyography of neck muscles | baseline and post- 4week intervention
  We will examine the value of Surface Electromyography of sternocleidomastoid muscle and upper trapezius muscle when they are cervical flexion, extension, flexion to the left and flexion to the right.
scores of the Neck Disability Index(NDI) | baseline and post- 4week intervention
  We will estimate the scores of NDI of participants.
scores of the Northwick Park Neck Pain Questionnaire (NPQ) | baseline and post- 4week intervention
  We will estimate the scores of NPQ of participants.
scores of Short-form McGill Pain Questionnaire(SF-MPQ) | baseline and post- 4week intervention
  We will estimate the scores of SF-MPQ of participants.

OTHER OUTCOMES:
degree of Evaluation of the therapeutic effect | baseline and post- 4week intervention
  We will estimate the degree of Evaluation of the therapeutic effect according to Standards of the diagnosis and the therapeutic effect of Disease and Syndrome of traditional Chinese medicine.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China